CLINICAL TRIAL: NCT06702865
Title: Combined Leadless Pacemaker and Left Atrial Appendage Occlusion Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tam Tsz Kin, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: LP LAAO registry
Record Dates: First submitted 2024-10-25; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Leadless Pacemaker; Left Atrial Appendage Occlusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- LP and LAAO: Patients indicated for combined leadless pacemaker and left atrial appendage occlusion will have combined procedure. Procedure will be performed with usual implantation techniques.

SUMMARY:
Leadless pacemakers (LP) are safe and effective alternatives to transvenous pacemakers in selected patients. Implantation is performed with a large caliber delivery catheter. Care must be taken in introducing the delivery catheter into the patient's venous system. Implantation in patients with small body habitus demands extra caution to avoid vascular injury and cardiac perforation. Negotiating the large caliber delivery catheter into the desired implant position may also be more difficult in small right ventricles. In a previous report of Micra leadless pacemakers, it was found that low BMI was associated with poor efficacy and safety.

The Aveir leadless pacemaker is a new leadless pacemaker that has obtained FDA approval and is commercially available in Hong Kong. It features a screw-in fixation mechanism, in contrast to the passive fixation of Micra. Most of its efficacy and safety data comes from a Western population. It would be important to study its efficacy and safety in an Asian population, who tend to have smaller body builds, hence more prone to complications.

In recent papers regarding the Micra leadless pacemaker, it was found that tricuspid regurgitation (TR) could be a result, especially if the implant was too close to the tricuspid valve. Given the almost 50% longer device dimension of the Aveir VR compared with the Micra leadless pacemaker (38mm vs 26mm), it is expected that the device mechanical interaction with tricuspid valve dysfunction can be more common. In the smaller hearts of an Asian population, it would be important to study the TR progression after device implantation.

About half of the patients implanted with leadless pacemakers were having concomitant atrial fibrillation and thus were at risk for thromboembolic events. Left atrial appendage occlusion was an effective procedure for stroke prevention in patients with atrial fibrillation. Because one patient often has indication for both LAAO and leadless pacemaker, combining them into the same procedure is appealing. The combined procedure can be performed with one single access. The imaging used to guide LAAO implantation can also be used to guide leadless pacemaker implantation to improve the procedure safety.

This study is a prospective observational study. Patients indicated for combined leadless pacemaker and left atrial appendage occlusion will be enrolled. Patients would fulfill guideline Class I and Class II indication for leadless pacemaker. The decision for left atrial appendage occlusion will be a shared decision-making process between the physician and patient. The consideration is usually based on patient's bleeding risk, tolerability for oral anticoagulation and patient preference.

DETAILED DESCRIPTION:
Baseline demographics will be collected, including body weight, body height, age, sex, comorbidities, indication of pacing and indication of left atrial appendage occlusion, etc.

Implantation of pacemaker will be performed with usual implantation techniques. During the implantation, procedural details will be collected. Any complications related to the implantation will be collected as well.

The implantation of LAAO will be performed with usual implantation techniques. Image guidance will be employed, such as transesophageal echocardiogram or intracardiac echocardiogram.

Patients will be followed up per routine clinical practice. During the clinical follow up, device measurements will be recorded. If any imaging is performed during follow up, the result will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18-year-old
2. Patients satisfying guideline Class I or Class II indication for pacemaker 6,7
3. Patients with atrial fibrillation
4. Patient deemed indicated for left atrial appendage occlusion after a shared decision making between physician and patient

Exclusion Criteria:

1. Pregnancy
2. Expected life expectancy <1 year
3. Patients with known mitral stenosis
4. LVEF <30%
5. Severe mitral regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient in Prince of Wales Hospital who is deemed indicated for left atrial appendage occlusion after a shared decision making between physician and patient
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Implant success rate | From implant to the date of study end, up to 12 months
  Evaluate implant success rate for both leadless pacemaker and left atrial appendage occlusion
Implant complications | From implant to the date of study end, up to 12 months
  Evaluate Implant complications

SECONDARY OUTCOMES:
Pacing parameters | From implant to the date of study end, up to 12 months
  Evaluate pacing parameters in follow up visits
Leadless pacemaker implantation locations | From implant to the date of study end, up to 12 months
  Evaluate implantation location of leadless pacemaker
Imaging | From implant to the date of study end, up to 12 months
  Follow up imaging results (CT or TEE) for leadless pacemaker and left atrial appendage occlusion
Rate of increase in tricuspid regurgitation severity | From implant to the date of study end, up to 12 months
  Evaluate rate of increase in tricuspid regurgitation severity by >=1 grade after leadless pacemaker implantation
Procedure time | On procedure date
  Evaluate the procedure time of combined procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong